CLINICAL TRIAL: NCT01759745
Title: The Influence of Gaze Shift and Emotions on Symptoms of Blepharospasm- a Pilot Study.
Brief Title: Influence of Gaze Shift and Emotions on Symptoms of Blepharospasm
Status: Withdrawn | Type: Observational
Why Stopped: Organisatory reason
Sponsor: Kirsten Elwischger, MD (Other)
Responsible Party: Sponsor-Investigator, Kirsten Elwischger, MD, Dr. Kirsten Elwischger, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: BEB_Gaze_Emotion
Record Dates: First submitted 2012-12-31; First posted 2013-01-03 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Pupillary Occlusion
MeSH Terms: conditions — Pupil Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blepharospasm: Blepharospasm, patient's group
- Control: Healthy control subjects

SUMMARY:
Blepharospasm (BEB) is a focal dystonia characterized by forceful, involuntary contractions of the orbicularis oculi muscle. (Jankovic et al 1983) Patients with BEB report task and situation specific modulations of their symptoms. So called "sensory tricks" are actions that minimize symptoms and include concentrating, talking, pulling on the eyelids, blowing air, and applying pressure to the periocular or temple region. (Weiner 1984) Many patients describe that other tasks/situations are exacerbate their symptoms specifically under bright fluorescent lights and stress. (Burke 1984) Earlier studies showed that blink patterns differ between BEB patients and control during rest, reading and talking.

In healthy subjects gaze evoked blinks are a physiologic phenomenon: initiation of gaze shifts evoke a blink, blinks facilitate gaze shifts. (Evinger 1994) In healthy subjects emotions and thoughts influence gaze shifts and blink rate. (Leal 2008, de Genaro 1988) However, little is known about various task and emotion specific influences on symptoms of BEB (e.g. expecting a gaze shift might worsen symptoms while driving a car).

Differences in emotion and gaze related blink patterns between patients and controls will contribute to the understanding of the pathophysiology of BEB. This might offer new therapeutic options, e.g. symptom modulation.

The investigators hypothesize that blink patterns, measured by duration and frequency of pupillary occlusion differ between patients and control, when performing gaze shifts and emotion related blink patterns, measured by duration and frequency of pupillary occlusion differ between patients and controls.

The aim of this pilot trial is to assess differences in gaze evoked and emotion related blink patterns between patients and controls. These differences might contribute to the understanding of the pathophysiology of BEB.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Willing to participate
* Idiopathic blepharospasm
* Age 18-80
* Last botulinum toxin injection <3months

Control:

* Willing to participate
* Age and sex matched with patients
* Age18-80

Exclusion Criteria:

Patients:

* Secondary blepharospasm
* Neurologic Comorbidities
* Other eye disease besides BEB
* History of neuroleptic medication
* Use of medications on the study day, that influence eye blinks& attention
* Drinking of caffeine or theine containing beverages on the study day

Patients and Control:

* Intake of psychotropic drugs at day of examination
* History of neuroleptic medication
* present eye disease
* Neurologic diseases that influence blinking
* Use of medications on the study day, that influence eye blinks& attention
* Drinking of caffeine or theine containing beverages on the study day

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 patients suffering from BEB, age 18-80 from our Botulinum toxin clinic will be investigated.
  For controls,20 healthy age matched subjects will be investigated. All participants will sign an informed consent.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-12 (Estimated); Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Duration and frequency of pupillary occlusion | At baseline
  Duration and frequency of pupillary occlusion during different tasks and situations will be studied via videooculography

SECONDARY OUTCOMES:
Number of blinks and spasms. | At baseline
  Number of blinks and spasms, registered by videotape of the eyes during different tasks and situations.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sycha, Prof.Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Neurology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Jankovic J, Ford J. Blepharospasm and orofacial-cervical dystonia: clinical and pharmacological findings in 100 patients. Ann Neurol. 1983 Apr;13(4):402-11. doi: 10.1002/ana.410130406. PMID 6838174
- [Background] Weiner WJ, Nora LM. "Trick" movements in facial dystonia. J Clin Psychiatry. 1984 Dec;45(12):519-21. PMID 6501239
- [Background] Burke RE, Fahn S, Marsden CD, Bressman SB, Moskowitz C, Friedman J. Validity and reliability of a rating scale for the primary torsion dystonias. Neurology. 1985 Jan;35(1):73-7. doi: 10.1212/wnl.35.1.73. PMID 3966004
- [Background] Richard MJ, Woodward DJ, McCoy AN, Woodward JA. Effect of reading on surface electromyogram recordings in patients with blepharospasm. Ophthalmic Plast Reconstr Surg. 2009 Sep-Oct;25(5):378-81. doi: 10.1097/IOP.0b013e3181b0d630. PMID 19966652
- [Background] Evinger C, Manning KA, Pellegrini JJ, Basso MA, Powers AS, Sibony PA. Not looking while leaping: the linkage of blinking and saccadic gaze shifts. Exp Brain Res. 1994;100(2):337-44. doi: 10.1007/BF00227203. PMID 7813670